CLINICAL TRIAL: NCT05419596
Title: The Analysis of Gene Variants Related to POCD in Elderly Patients: a Prospective, Observational Study
Brief Title: The Analysis of Gene Variants Related to POCD in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Other Study IDs: 2022/711
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Urologic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be evaluated using DNA sequence analysis, Realtime PCR, and ELISA techniques. Proteins including APOE, phosphatidyl inositol-binding clathrin assembly protein, CR1 - complement receptor 1, ATP-binding cassette transporter, IL6,Triggering receptor expressed on myeloid cells2 (TREM2) will be investigated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major Urologic Surgery Group: Elder patients who undergo major urologic surgery will be investigated for the change in genomic protein that are related to cognition. These proteins are APOE, phosphatidyl-inositol-binding clathrin assembly protein, CR1 (complement receptor 1) , ATP-binding cassette transporter, IL6, Triggering receptor expressed on myeloid cells2 (TREM2)
  Interventions: Procedure: Urologic Surgery

INTERVENTIONS:
Procedure: Urologic Surgery — Patients undergoing major urologic surgery will be examined with blood samples that will be taken preoperatively and postoperatively. Accordingly several gene variants and proteins will be examined for patients with or without postoperative cognitive dysfunction. These proteins consist of APOE, phosphatidyl-inositol-binding clathrin assembly protein, CR1 - complement receptor 1 , ATP-binding cassette transporter, IL6, Triggering receptor expressed on myeloid cells2 (TREM2).

SUMMARY:
The pathophysiology of postoperative cognitive dysfunction (POCD) following surgery may be related to Alzheimer's disease. Different studies show that; low levels of glial cell line-derived growth factor are found in both POCD and Alzheimer, and brain cholinergic markers like Choline acetyl transferase activity, High affinity choline uptake activity, and Acetil Choline (Ach) activity are decreased in Alzheimer disease.We know cholinergic inputs in the basal forebrain have a critical role in many other functions including memory, attention, arousal and sensory processing.

Cholinergic neuron located basal section of forebrain degenerate extensively in Alzheimer disease which shares similarities with postoperative delirium and POCD. Ach binds to two well-known receptors in brain that are Nicotinic receptors which implicate several important functions such as "memory, learning, arousal and reward" and Muscarinic receptors which are widely distributed in forebrain and play an important role of development delirium and POCD. Dysfunction of cholinergic system may be one key aspect of postoperative DELIRIUM, POCD and ALZHEIMER disease.

In this investigation; we would like to evaluate the relationship between genes encoding inflammation-related mediators detected in postoperative cognitive dysfunction and gene variants in Alzheimer's disease in a larger panel for elder patients undergoing major urologic surgery. Therefore our study will focus on demographic information of the patients (age, gender, comorbidity), neurocognitive tests (1 week before the surgery, postoperative 1st week and postoperative 3rd month), intraoperative data (mean arterial pressure, heart rate, need for inotrope, duration of mechanical ventilation, need for transfusion), and biochemical tests (Preoperative and postoperative blood samples for each patient) which are APOE, phosphatidylinositol-binding clathrin assembly protein, CR1 - complement receptor 1, ATP-binding cassette transporter, IL6, TREM.

ELIGIBILITY:
Inclusion Criteria:

* Patients over age of 60 years
* Patients scheduled for major urologic surgery

Exclusion Criteria:

* Failure of the patient or the person with legal authority to make a decision about him/her.
* Patients with severe hearing-vision problems before surgery.
* Patients with severe neurological-psychiatric disorders before surgery.
* Patients who cannot find a common language.
* Emergency surgeries

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are over 60 years old and scheduled for elective/semielective major urologic surgery
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-25 (Estimated)

PRIMARY OUTCOMES:
Change in Interleukin-6 levels in elder atients undergoing major urologic surgery | From preoperative 1 hour to postoperative 2 hours
  Major urologic surgery patients will be evaluated for their different genomic protein levels that are possibly related to cognitive disorders. These proteins consist of APOE, phosphatidylinositol-binding clathrin assembly protein, CR1 (complement receptor 1) , ATP-binding cassette transporter, Interleukin- 6, Triggering receptor expressed on myeloid cells2 (TREM2). Accordingly two blood samples will be gathered from each patient in the preoperative and postoperative period.

SECONDARY OUTCOMES:
Addenbrooke cognitive examinations change (Preoperative to postoperative) | Up to Postoperative 7 days.
  Addenbrooke test will be applied the day before the surgery (T1) and 7 days after the surgery (T2). 0 reflecting the worst and 100 reflecting the best values, 1 standart deviation worsening between the tests will be accepted as Postoperative Cognitive Dysfunction (POCD). Patients with POCD will be accepted as Group POCD (+), without POCD will be accepted as Group POCD (-)
Addenbrooke cognitive examinations change for the chronic period | Up to postoperative three months
  Third Addenbrooke test will be applied on the postoperative third month (T3). Difference between T3 and T2 will be recorded
The difference in IL-6 between the groups | Up to postoperative 1 hour
  Postoperative IL-6 level difference in Group POCD (+) versus Group POCD (-).
DNA sequence analysis of APOE gene | Up to postoperative 1 hour
  DNA sequence analysis of APOE in whole patient group.
DNA sequence analaysis of phospatydil-inositol binding clathrin gene | Up to postoperative 1 hour
  DNA sequence analaysis of phospatydil-inositol binding clathrin gene in whole patient group
DNA sequence analysis of complement receptor 1 protein gene | Up to postoperative 1 hour
  DNA sequence analaysis of complement receptor 1 protein gene in whole patient group
DNA sequence analysis of Triggering receptor expressed on myeloid cells2 (TREM2) | Up to postoperative 1 hour
  DNA sequence analysis of Triggering receptor expressed on myeloid cells2 (TREM2) in whole patient group
DNA sequence analysis of ATP-binding cassette transporter gene | Up to postoperative 1 hour
  DNA sequence analysis of ATP-binding cassette transporter gene in whole patient group